CLINICAL TRIAL: NCT05308745
Title: The Effects of a Probiotic Milk Drink, Yakult®, Containing Lactobacillus Casei Shirota on the Intestinal Microbiota and Intestinal Environment in Residents and Staff at Elderly Houses in Indonesia
Brief Title: Effects of Yakult Ingestion in Residents and Staffs at Indonesian Elderly Houses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endang Sutriswati Rahayu (Other)
Collaborators: Yakult Honsha Co., LTD (Industry)
Responsible Party: Sponsor-Investigator, Endang Sutriswati Rahayu, Prof. Dr. Ir., Gadjah Mada University
Organization: Gadjah Mada University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YH.03.2018
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: probiotic; elderly subject; intestinal microbiota

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic group (Active Comparator): Participants within this group consumed Yakult® as research product 1 bottle/day for 24 weeks (168 days).
  Interventions: Dietary Supplement: Yakult®
- Placebo group (Placebo Comparator): Participants within this group consumed placebo as research product 1 bottle/day for 24 weeks (168 days).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Yakult® — Fermented milk drink containing over 6.5×10^9 CFUs of L. casei Shirota/65 ml
  Arms: Probiotic group
Dietary Supplement: Placebo — Taste, appearance, component, and number of calories are the same as Yakult®, non-fermented milk product
  Arms: Placebo group

SUMMARY:
A study to investigate the effect of Yakult® containing L. casei Shirota on the intestinal microbiota, intestinal environment, and stool frequency in healthy adult and elderly subjects in Indonesia. The clinical phase of this study was conducted for 26 weeks in three different elderly houses. The subjects were grouped into two categories: probiotic and placebo group, according whether the subjects consumed product or placebo samples. Fecal sampling were taken three times during the study.

DETAILED DESCRIPTION:
The study investigates the ingestion effect of a commercialized probiotic milk drink, Yakult®, for residents and staffs at Indonesian elderly houses (age limit: 18 - 95 years old). The study will be conducted as a double blind, placebo controlled parallel comparison study. There will be 26 weeks used for the study, comprised of: A 2-week baseline assessment period, and 24-week probiotic or placebo intake period.

From 112 subjects, the participants will be grouped into two: probiotic and placebo group. Those in probiotic group will consume Yakult® (Fermented milk drink containing over 6.5×10^9 CFUs of L. casei Shirota/65 ml), while placebo group will consume the placebo product (taste, appearance, component, and number of calories are the same as Yakult®, non-fermented milk product). The treatment intake will be done for 24 weeks (182 days).

During the study, the participants are expected to fill questionnaire of frequency of bowel movements and Chinese Constipation Questionnaire to obtain the defecation frequency (Bristol Stool score) and abdominal symptom scores. Fecal samples will be collected three times: on the last day of the baseline period (day 14±1), 12 weeks (day 98±1) after intake period, after the 24-weeks intake period (day 182±1). Afterwards, the obtained fecal samples will be further analyzed for its microbial composition, level of short-chain fatty acids and putrefactive compounds.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign written informed consent
* Healthy adult and elderly subjects (adult: between 18 - 69 years old; elderly at least 70 years old.
* No history of an adverse reaction to any of the components of the active or placebo versions of the probiotic product.
* Can eat, regularly.
* Has been diagnosed by doctors as healthy both physically and mentally.
* Can abide by the experimental protocol.

Exclusion Criteria:

* Excessive alcohol consumption (defined as follows: male; over 28 glasses a week, female; over 21 glasses/week).
* Consume antibiotics or laxatives at least 2-week prior screening period.
* Consume ingestion of fermented dairy foods (yogurt), probiotic foods and/or prebiotic at least 2 weeks prior to the study.
* Reported current usage of Narcotics and Psychotropic,
* History of GI surgery i.e. Colectomy and Enterectomy.
* Symptoms meeting to Rome IV diagnostic criteria for irritable bowel syndrome
* Pregnant or childbearing women

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Beneficial impact of Yakult on intestinal microbiota and intestinal environment compared to Placebo | up to 23 months
  Fecal samples will be analyzed for its microbiota composition using YIF-SCAN (Yakult Intestinal Flora Scan) and 16S rRNA gene sequencing will be utilized to measure the intestinal microbiota. The basic principle of YIF-SCAN is the quantitative RT-PCR method. The microbiota composition that will be analyzed is the number and ratio of beneficial bacteria (ex. Bifidobacterium) and harmful bacteria (Enterobacteriaceae, Enterococcus, C. perfringens, C. difficile etc.)

SECONDARY OUTCOMES:
Frequency of bowel movements | up to 23 months
  Using the Bristol Stool scale and stool frequency questionnaire, the frequency of bowel movements are measured as Bristol Stool score
Abdominal symptom scores | up to 23 months
  Using the Chinese Constipation questionnaire, bowel function and rectal symptoms are documented
The concentration of total short chain fatty acids | up to 23 months
  The level of several short-chain fatty acids are measured from stool samples. These fatty acids are acetic acid, propionic acid, butyric acid, iso-butyric acid, succinic acid, lactic acid, formic acid, iso-valeric acid, valeric acid
The contents of putrefactive production | up to 23 months
  The concentration of several putrefactive compounds are measured from stool samples. These compounds include ammonia, phenol, indole, p-cresol.

CONTACTS AND LOCATIONS:
Overall Officials: Endang Sutriswati Rahayu, Principal Investigator — Gadjah Mada University
Locations (3):
- Indonesia (3):
  - Wana Seraya Elderly House, Denpasar, Badung
  - Tresna Werda Jara Mara Pati Elderly House, Singaraja, Buleleng
  - Werdha Santi Elderly House, Tabanan